CLINICAL TRIAL: NCT04188743
Title: DEKODON: Decolonization of Gram-negative Multi-resistant Organisms (MDRO) with Donor Microbiota (FMT)
Brief Title: Decolonization of Gram-negative Multi-resistant Organisms (MDRO) with Donor Microbiota (FMT)
Acronym: DEKODON
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC-3034; 2018/0966 (Other: EC UZG)
Record Dates: First submitted 2019-10-17; First posted 2019-12-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Resistance Bacterial
Keywords: Fecal Microbiota Transplantation; Hospitals, Isolation; Drug Resistance, Multiple, Bacterial; Gram-Negative Bacteria; Gastrointestinal Microbiome
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: 150 participants will be randomly allocated to an "intervention" group (100p) and a "no intervention" group (50p). Participants in the "intervention" group will be randomised (double blind) to either fecal microbiota transfer with donor stool (allogenic FMT) or fecal microbiota transfer with own stool (autologous FMT). Participants in the "no intervention" group will be monitored without receiving a fecal microbiota transfer.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Allogenic FMT (Experimental): Participants in the allogenic FMT- group will receive FMT-treatment using healthy donor microbiota supplied by the Ghent Stool Bank. The donor stool (50g) is processed shortly after production and tested intensively. It's frozen at -80°C until administration via naso-duodenal/-jejunal tube (Cortrak).
  Interventions: Biological: Allogenic FMT
- Autologous FMT (Placebo Comparator): Participants in the autologous FMT- group will receive FMT-treatment using their own microbiota to account for effects due to the treatment itself. Their stool is processed as close to the treatment as feasible. It's processed and frozen at -80°C until administration via naso-duodenal/-jejunal tube (Cortrak).
  Interventions: Biological: Autologous FMT
- No intervention (No Intervention): Participants in the "No intervention"-group will not receive any treatment but will be monitored similarly as the "Allogenic FMT" and "Autologous FMT" groups.

INTERVENTIONS:
Biological: Allogenic FMT — Transplantation of fecal microbiota from a donor into a recipient
  Other Names: Fecal Microbiota Transplantation with donor stool; Fecal Microbiota Transfer with donor stool
  Arms: Allogenic FMT
Biological: Autologous FMT — Transplantation of autologous fecal microbiota
  Other Names: Fecal Microbiota Transplantation with own stool; Fecal Microbiota Transfer with own stool
  Arms: Autologous FMT

SUMMARY:
Colonization by Multiple Drug Resistant Organisms (MDROs) during patient hospitalization requires expensive isolation measures and renders the return or transfer to other departments or institutions often impossible. Currently there is no specific treatment available. Patients have to wait for spontaneous clearance which can take months or does not happen at all.

The study will test the effect of Fecal Microbiota Transfer (FMT) on gut MDRO colonization. The focus will be on patients with a long-term colonization by Gram-negative bacteria for which isolation is warranted. Participants will be randomized into two treatment groups; allogenic FMT versus autologous FMT. A third group of participants will be monitored but will not receive an FMT. Decolonization rate will be compared one month after treatment. Additionally gut microbial composition will be studied up to one year after FMT.

DETAILED DESCRIPTION:
This double-blind controlled randomized study will test the efficacy of Fecal Microbiota Transfer (FMT) on gut Multiple Drug Resistant Organism (MDRO) colonization.

Participants:

The study targets hospitalized patients (>18 years old) that need to stay in isolation because of colonization by Carbapenem-resistant Enterobacteriales (CRE), non-E. coli Enterobacteriales that produce extended spectrum beta-lactamase (ESBL) or Multi Drug Resistant (MDR) Pseudomonas and MDR Acinetobacter species. Participants will be randomized in two groups (allogenic and autologous FMT). Additionally a third group of participants will be monitored without intervention.

Treatment:

Participants in the allogenic FMT- group will receive treatment using healthy donor microbiota preferably through naso-duodenal/-jejunal administration (Cortrak). Donor material will be supplied by the Ghent Stool Bank. The colonization status will be monitored on a regular basis (at least once per week) by culturing fecal swabs. Additionally fecal samples will be taken on fixed time points for microbial composition analysis (16S ribosomal ribonucleic acid metagenomics).

Controls:

Participants in the autologous FMT-group will will receive an FMT with their own microbiota to account for the effects of the intervention itself. Participants in the "no intervention" group will not receive an FMT. Both control groups will be monitored and sampled identically to the allogenic FMT-group.

Outcome:

The primary outcome (MDRO-decolonization rate in treatment versus control) will be evaluated 1 month after FMT. Secondarily, safety and tolerability of the treatment will be assessed. The patients will be monitored up to 1 year after treatment to evaluate microbiome composition and to define parameters in the microbiome that are associated with clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age, and must sign the 'informed consent' form and thus agree with the data collection, sampling and FMT.
* At least 2 consecutive confirmations of MDRO colonization in faeces, which complicate the necessary follow-up and/or therapy for the patient.
* Participants must be able to endure the treatment (evaluated by treating physician).

Exclusion Criteria:

* Inflammatory bowel disease (Crohn's disease, ulcerative colitis ...)
* Diagnosed hereditary blood disease (Haemophilia, Von Willebrand ...)
* Chronic liver disease
* Active drug use or alcohol abuse / dependence, which according to the researchers' opinion may interfere with the patient's participation in the study
* Simultaneous use of probiotics (except yoghurt)
* Existing immune deficiency (congenital or acquired), or concomitant immunomodulatory treatment (including systemic corticosteroids) in the 12 weeks prior to randomization, nasal or inhaled corticosteroid use is permitted
* Positive pregnancy test (or potentially pregnant)
* Breastfeeding
* Severe food allergy (anaphylaxis, urticarial)
* Antibiotic treatment up to 7 days before FMT, or planned to start within one month after FMT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with decolonization success/failure | 1 month after treatment
  These participants were screened positive for MDRO's in stool cultures before treatment and monitored at least once per week up to 1 month after treatment. "Decolonization" = 3 consecutive negative cultures in minimal time span of 2 weeks.

SECONDARY OUTCOMES:
Side effects | up to 1 year after treatment
  Monitor adverse events
Treatment effect on microbial community in participants | up to 1 year after treatment
  Evaluation of gut bacterial composition changes in participants over time pre- and post-treatment with 16S ribosomal ribonucleic acid based metagenomic analysis.
Treatment tolerability | 1 month after treatment
  The tolerability of the treatment is monitored with an in-house developed questionnaire considering the participant's opinion before, during and after the treatment on a score of 1 (very bad) to 5 (very good).

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Verhasselt, Prof. Dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be pseudonymized, not traceable to participant identity except for clinical staff. All participant data, questionnaires, colonization and sequencing data annotation will be collected in "open REDCap" (TLS encrypted secure web platform) to ensure traceability and safekeeping of the data. Data is stored and backed-up for at least 20 years on a secured server.
  Following data will be shared with other researchers:
  * baseline characteristics (age, BMI, sex...)
  * colonization status
  * analyzed gut microbial sequencing data
  * clinical follow-up data
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of the primary publication